CLINICAL TRIAL: NCT02598219
Title: Randomized Trial Comparing Sentinel Node (SN) Policy to Current French Initial Staging Protocols in Early Stage Endometrial Carcinomas at Intermediate and High Risk of Recurrence
Brief Title: Evaluation of Sentinel Node Policy in Early Stage Endometrial Carcinomas at Intermediate and High Risk of Recurrence.
Acronym: SENTIRAD
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: National Cancer Institute, France (Other Government); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Canceropôle Nord Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SENTIRAD-1502
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Non Endometrioid Carcinoma; Endometrioid Carcinoma
Keywords: Sentinel node
MeSH Terms: conditions — Carcinoma, Endometrioid | interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-operative SN mapping with radionucleide (Experimental): 1 Pre-operative Sentinel Node (SN) mapping with Nanocis or Nanocoll or Rotop-nanoHSA
  2- Intra-operative SN mapping with patent V blue dye, or Intra-operative SN mapping with indocyanin green for patients with known hypersensitivity, allergy to patent V blue dye
  3- Full bilateral laparoscopic lymphadenectomy and Hysterectomy: If bilateral SN are detected, all positive SN are removed, then the surgeon proceeds to a total hysterectomy.
  If unilateral SN are detected, surgeon will complete intervention with pelvic LN dissection on the opposite side, in accordance with risk group definition (ex: omentectomy for high-risk non endometrioid carcinomas).
  If non SN are detected, surgeon will proceed to a total hysterectomy, a bilateral salpingo-oophorectomy, a complete and bilateral pelvic LND with more enlarged dissection regardless the pathology
  Interventions: Drug: Pre-operative SN mapping with radionucleide; Drug: Intra-operative SN mapping with patent V blue dye; Drug: Intra-operative SN mapping with indocyanin green; Procedure: Full bilateral laparoscopic lymphadenectomy and Hysterectomy
- B : Current initial staging protocols (Other): Current initial staging protocols
  Interventions: Procedure: Current initial staging protocols

INTERVENTIONS:
Drug: Pre-operative SN mapping with radionucleide — 1. Preparation : four 1ml syringe (Nanocis, or Nanocoll, or Rotop-nanoHSA) are prepared per patient, each containing a total activity 10 MBq if the injection is planned the same day of surgery and in the operative theater OR each containing a total activity 30MBq if the injection is performed the day before the surgery.
  2. Intracervical injection is performed by the surgeon, no more than 3-24 hours before surgery : 4 submucous injections with the filtered radiocolloid at 3, 6, 9 and 12 o'clock positions. Each injection if performed at 2 mm of depth for a total activity of 40 MBq or a total activity of 120 MBq is the surgery is planned the day after the injection.
  3. Sentinel Node detection by planar scintigraphy at 1 and 3h (if no detection at 1 hour), or by SPECT-CT imaging if available.
  Other Names: Pre-operative Sentinel Node
  Arms: Pre-operative SN mapping with radionucleide
Drug: Intra-operative SN mapping with patent V blue dye — 1. Patent blue V dye are diluted with saline sterile solution to obtain 4ml of 50%. Four 1ml syringe, each containing a 50% patent blue dye solution, are prepared per patient.
  2. Intracervical injection is performed by the surgeon. after anesthesis induction and incising the skin,under laparoscopic / laparotomy control to detect intraperitoneal injection of the tracer. Sub-mucous injections are performed with 50% diluted dye at 3 and 9 o'clock positions. At each positions : 1ml is injected deep into the stroma of the cervix (1cm), another 1ml is injected superficially (at 2mm depth). The time between the injection of the dye and the search for the SN must be as shortest as possible.
  3. SN are detected by direct visualization of blue colored lymphatics and node
  Other Names: Intra-operative SN mapping
  Arms: Pre-operative SN mapping with radionucleide
Drug: Intra-operative SN mapping with indocyanin green — 1: Infracyanine powder is diluted in aqueous sterile water to obtain 4ml with a concentration of 1.25 mg/mL. Four 1ml syringe, each containing a 1.25 mg/mL Infracyanine dye solution, are prepared per patient.
  2- Intracervical injection is performed by the surgeon, after anesthesis induction and incising the skin,under laparoscopic / laparotomy control to detect intraperitoneal injection of the tracer. Sub-mucous injections are performed with 50% diluted dye at 3 and 9 o'clock positions. At each positions : 1ml is injected deep into the stroma of the cervix (1cm), another 1ml is injected superficially (at 2mm depth). The time between the injection of the dye and the search for the SN must be as shortest as possible
  3- SN detection by near-infrared fluorescence imaging
  Other Names: Intra-operative Sentinel Node (SN) mapping with Infracyanine
  Arms: Pre-operative SN mapping with radionucleide
Procedure: Full bilateral laparoscopic lymphadenectomy and Hysterectomy — * Bilateral pelvic lymphadenectomy (intermediate risk endometrioid)
  * Or Ilio-infrarenal paraaortic lymphadenectomy (high risk endometrioid)
  * Or Pelvic + paraaortic lymphadenectomies (high risk non endometrioid)
  Other Names: Full bilateral lymphadenectomy
  Arms: Pre-operative SN mapping with radionucleide
Procedure: Current initial staging protocols — Current French initial staging protocols
  Arms: B : Current initial staging protocols

SUMMARY:
The aim of this trial is to evaluate the sentinel node policy in early stage endometrial carcinomas at intermediate and high risk of recurrence (by comparing the sentinel node policy to current initial staging protocols).

DETAILED DESCRIPTION:
1. Routine exams required for diagnosis:

   * Endometrioid biopsy or product of a dilatation-curettage under hysteroscopy for diagnosis of histologic typing
   * Tumor assessment: Lombopelvic MRI (1.5 or 3T) with gadolinium injection, studied by steady and dynamic sequences. US and CT-Scan in case of intolerance to MRI should be discussed. FDG-PET may be an option.
2. Tumor board: The completed chart will be reviewed to confirm the risk group and indication.
3. Complete physical and gynecological examination by surgical oncologist followed by a consultation of anesthesiology to confirm the operability of patient.
4. Informed and signed consent form.
5. Study baseline assessment.

   Then,
6. Surgery should be performed within a maximum of 4 weeks from the first consultation, according arm allocated:

   Arm A: Sentinel node policy*

   Arm B:
   * Bilateral pelvic lymphadenectomy (intermediate risk endometrioid)
   * Or Ilio-infrarenal paraaortic lymphadenectomy (high risk endometrioid)
   * Or Pelvic + paraaortic lymphadenectomies (high risk non endometrioid)*

     * along with a peritoneal staging for each arm (cytology, random biopsies, infracolic omentectomy)
7. Second tumor board: after definitive pathological results of the hysterectomy-annexectomy and node (sentinel or not) specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with early endometrial carcinoma with early FIGO clinical stage I-II (clinical examination, abdomino-pelvic MRI/Ultrasound - or CT scan if MRI not possible - and endometrial biopsy or curettage), then stratification of the recurrence risk as defined by last European Society for Medical Oncology (ESMO) guidelines :

   * Intermediate-risk endometrioid (type 1): FIGO stage IA/T1a grade 3, or IB grade 1 or 2
   * Or High risk endometrioid (type 1) : FIGO stage IB/T1b grade 3, or II grade 1 or 2 or 3
   * Or High risk non endometrioid (type 2) : FIGO stages I-II
2. Without any suspicious pelvic, paraaortic, distant node at preoperative MRI
3. Age ≥ 18 years
4. Performance status (OMS) ≤ 2
5. No contraindication to surgery
6. Absence of known hypersensitivity to colloidal rhenium sulphide and technetium (nanocolloid) or one of its excipients, to human albumin preparations, to Nanocoll® and Rotop-nanoHSA® and their excipients, to injectable dyes (blue dye or indocyanine green if available) or one of their excipients, to triphenylmethane derivatives
7. Signed and dated informed consent
8. Effective contraception for patients with reproductive potential
9. Patient affiliated with a health insurance system

Exclusion Criteria:

1. Preoperative workup with :

   * Previous hysterectomy (by nature, this trial cannot be offered as a secondary staging procedure)
   * non carcinoma (for example sarcoma, trophoblastic tumor)
   * Low-risk endometrioid carcinoma as defined by the ESMO: 2009 FIGO stage IA grade 1-2
   * Metastatic disease at preoperative workup
   * Suspicious adenopathy at preoperative workup
2. Pregnant and/or breastfeeding woman
3. No understanding of the trial
4. Patient deprived of liberty or in guardianship
5. Inexperience of the trial site in pelvic sentinel node detection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2024-10 (Actual); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Morbidity | Up to 3 after surgery
  Per-operative morbidity will be assessed during surgery according to the Oslo classification of intraoperative unfavourable incidents.
  Early post-operative morbidity will be assessed up to 30 days and scored according to Clavien-Dindo scale. Distant complications, beyond day 30 for patients with no indication of a secondary surgical staging (e.g. secondary paraaortic dissection for pelvic pN1) will be evaluated in accordance with the NCI-CTCAE scale v4.03

SECONDARY OUTCOMES:
Rate of detected sentinel node | During surgery
  number of patients with ≥ 1 Sentinel Node (SN) / total number of explored patients, and bilaterality
Rate of pN1 | an average of 1 month after surgery
  n pN1 / total N
Disease free survival | Up to 5 years after surgery
  Time from the date of randomization to the first documentation of local, regional or distant disease or death, whichever occurs first.
Overall survival | Up to 5 years after surgery
  Time from the date of randomization to the date of death (indicate if the death is due to disease progression or not).
Pronostic value of L1CAM on the risk of reccurrence | an average of 1 month after surgery
  A standard staining with HES is carried out in a systematic manner as well as immunohistochemistry with polyclonal anti-L1CAM. If 10% or more of the tumor cells showed L1CAM staining, the sample is rated positive. The rate of L1CAM positive sample will be further correlated with the node involvement and disease recurrence.
Proteomic signature of positive SN | an average of 1 year after surgery
  Detection of SN involvement with proteomics

CONTACTS AND LOCATIONS:
Overall Officials: Lucie BRESSON, MD, Study Director — Centre Oscar Lambret
Locations (16):
- France (16):
  - Polyclinique Urbain V, Avignon
  - Centre Hospitalier Régional Universitaire, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Hôpital Jeanne de Flandres, CHRU Lille, Lille
  - Hôpital Mère-Enfant, CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Hôpital La Pitié-Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Institut de Cancérologie de l'Ouest, René Gauducheau, Saint-Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aboulouard S, Wisztorski M, Duhamel M, Saudemont P, Cardon T, Narducci F, Lemaire AS, Kobeissy F, Leblanc E, Fournier I, Salzet M. In-depth proteomics analysis of sentinel lymph nodes from individuals with endometrial cancer. Cell Rep Med. 2021 Jun 15;2(6):100318. doi: 10.1016/j.xcrm.2021.100318. eCollection 2021 Jun 15. PMID 34195683
- See also: Results of proteomics profiling of sentinel lymph nodes — https://pubmed.ncbi.nlm.nih.gov/34195683/